CLINICAL TRIAL: NCT06366789
Title: A Phase 1, Open-label, Dose Escalation and Dose Expansion, Multicenter Clinical Trial to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of ZE46-0134 in Adults With FLT3 Mutated or Spliceosome Mutated Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Dose Escalation and Expansion Study to Evaluate the Safety, PK, PD and Efficacy of ZE46-0134 in Adults With FLT3 Mutated or Spliceosome Mutated Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lomond Therapeutics Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZE46-0134-0002; CT-2024-CTN-00161-1 (Other: Therapeutic Goods Administration)
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: AML With Gene Mutations

STUDY DESIGN:
Intervention Model Description: dose escalation and dose optimization study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- ZE46-0134 Dose Level -1 (Experimental): Optional and would only be performed Dose Level 1 is poorly tolerated
  Interventions: Drug: ZE46-0134
- ZE46-0134 Dose Level 1 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE46-0134 Dose Level 2 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE46-0134 Dose Level 3 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE46-0134 Dose Level 4 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE46-0134 Dose Level 5 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE46-0134 Selected dose 1 (Experimental): The doses used in Part 2 of the study will be determined based on the data from Part 1 of the study and will not exceed a loading dose of 150 mg x 2 days and maintenance dose of 50 mg QD
  Interventions: Drug: ZE46-0134
- ZE46-0134 Selected dose 2 (Experimental): The doses used in Part 2 of the study will be determined based on the data from Part 1 of the study and will not exceed a loading dose of 150 mg x 2 days and maintenance dose of 50 mg QD
  Interventions: Drug: ZE46-0134
- ZE46-0134 Dose Level 6 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE46-0134 Dose Level 7 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE46-0134 Dose Level 8 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE50-0134 (Group 2) Dose Level -1 (Experimental): Optional and would only be performed Dose Level 1 is poorly tolerated
  Interventions: Drug: ZE46-0134
- ZE50-0134 (Group 2) Dose Level 1 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE50-0134 (Group 2) Dose Level 2 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE50-0134 (Group 2) Dose Level 3 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE50-0134 (Group 2) Dose Level 4 (Experimental)
  Interventions: Drug: ZE46-0134
- ZE50-0134 (Group 2) Selected dose 1 (Experimental): The doses used in Part 2 of the study will be determined based on the data from Part 1 of the study.
  Interventions: Drug: ZE46-0134
- ZE50-0134 (Group 2) Selected dose 2 (Experimental): The doses used in Part 2 of the study will be determined based on the data from Part 1 of the study.
  Interventions: Drug: ZE46-0134

INTERVENTIONS:
Drug: ZE46-0134 — oral capsules QD

SUMMARY:
This is a clinical study aiming to assess pharmacokinetics, pharmacodynamics and preliminary efficacy of ZE46-0134 in patients with FLT3 and spliceosome mutated Relapsed or Refractory Acute Myeloid Leukemia

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multicenter, dose escalation, and dose optimization study to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of ZE46-0134 in adult patients with relapsed or refractory AML with FLT3-ITD and/or FLT3-TKD mutations and spliceosome mutations. Patients with AML that are out-patients or hospitalized due to their AML can be enrolled in the study.

The study will be run in 2 parts: Part 1 will be dose escalation and determination of MTD, and Part 2 will be dose expansion.

Part 1 of the study will have 2 groups. Group 1: 3 to 6 eligible patients with FLT3 mutation will be sequentially enrolled into each of 8 planned dose level cohorts. Patients will receive up to 24 cycles (28 days each) of study treatment. For patients that continued to derive benefit after 24 cycles of treatment, continuation of ZE46-0134 therapy will be considered. Group 2: 3 to 6 eligible patients with spliceosome mutation will be sequentially enrolled into each of 4 planned dose level cohorts. Patients will receive up to 24 cycles (28 days each) of study treatment. For patients that continued to derive benefit after 24 cycles of treatment, continuation of ZE46-0134 therapy will be considered.

In Part 2, the dose expansion phase will involve enrolling up to 30 patients across 2 dose cohorts (i.e., 15 patients per cohort) for Group 1 and up to 30 patients across 2 dose cohorts (i.e., 15 patients per cohort) for Group 2. ZE46-0134 will be dosed as described for Part 1 of the study. The doses used in Part 2 of the study will be determined based on the data from Part 1 of the study.

Indication background information:

Acute myeloid leukemia (AML) comprises a heterogeneous group of aggressive blood cell cancers that arise from clonal expansion of malignant hematopoietic precursor cells in the bone marrow (BM) and is the most commonly diagnosed adult leukemia with a median age at diagnosis is 68 years, with an overall survival (OS) rate of 29.8%. As patients age, there is a 10% decrease in 5-year OS for every additional decade of life, with a 5-year OS of 0.4% in patients age >85 years1. Furthermore, remission rates and OS depend on a number of other factors, including cytogenetics, previous BM disorders, and comorbidities.

FMS-like tyrosine kinase-3 (FLT3) is a receptor tyrosine kinase (RTK) primarily expressed on immature hematopoietic progenitors and hematopoietic stem cells. FLT3 signaling is initiated when FLT3 ligand binds to FLT3, inducing the dimerization and activation of FLT3 via autophosphorylation. This then activates downstream signaling of phosphoinositide 3-kinase/protein kinase B (PI3K/PKB), mitogen-activated protein kinase (MAPK), and JAK2/STAT5 which leads to cell proliferation and suppression of apoptosis2.

FLT3 kinase is directly implicated in the pathogenesis of hematologic malignancies, particularly AML. FLT3 mutations are the most frequently identified mutations in AML patients. Activating mutations in FLT3, which are FLT3-internal tandom duplication (ITD) and FLT3 tyrosine kinase domain (TKD) mutations, account for 30% of all AML cases2. As a result of these mutations, the FLT3 receptor is continuously activated leading to the continuous activation of downstream signaling pathways, PI3K/AKT, MAPK, and signal transducer and activator of transcription (STAT5), resulting in increased cell proliferation and decreased apoptosis.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent must be obtained from the patient or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
2. Patient is ≥18 years of age at the time of obtaining informed consent.
3. Patient is refractory to or relapsed after first-line AML therapy (with or without HSCT).
4. Group 1: Patient must have a confirmed FLT3-ITD or FLT3-TKD mutation by central laboratory testing. Group 2: Patient must have a documented SF3B1, SRSF2, U2AF1, or ZRSR2 pathogenic mutation by local lab sequencing.
5. For Group 1 only: Patients must have previously been treated with Gilteritinib with failure to stop disease progression, or not met the criteria for treatment with Gilteritinib in the opinion of the Investigator, or chosen not to have treatment with Gilteritinib for social reasons.
6. Patients have a life expectancy of at least 3 months in the opinion of the Investigator.
7. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
8. Patient must meet the following criteria as indicated on the clinical laboratory tests:

   1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN)
   2. Serum total bilirubin ≤1.5 × ULN unless due to Gilbert's disease
   3. Estimated glomerular filtration (eGFR) rate of >50 mL/min as calculated by the Modification of Diet in Renal Disease equation.
9. Female patients:

   1. If of non-childbearing potential i.e., surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 6 weeks before the Screening visit or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone (FSH) level consistent with postmenopausal status, per local laboratory guidelines), or
   2. If of childbearing potential, must:

   i. Have a negative serum pregnancy test at the Screening visit and urine pregnancy test on admission to the clinic on Day-1.

   ii. Agree not to attempt to become pregnant or donate ova from signing the consent form until at least 45 days after the last dose of study drug.

   iii. Agree to use adequate contraception (defined as use of a condom by the male partner combined with use of a highly effective method of contraception from Screening until at least 45 days after the last dose of study drug, if not exclusively in a same-sex relationship or abstinent as a committed lifestyle).
10. Male patients and their female spouse/partners who are of childbearing potential must agree to use highly effective contraception consisting of 2 forms of birth control (at least 1of which must be a barrier method) starting at Screening and continue throughout the study period and for 45 days after the final study drug administration. Male patient must not donate sperm starting at Screening and throughout the study period and for 45 days after the final study drug administration.

Exclusion Criteria:

1. Written Informed Consent must be obtained from the patient or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
2. Patient is ≥18 years of age at the time of obtaining informed consent.
3. Patient is refractory to or relapsed after first-line AML therapy (with or without HSCT).
4. Patient must have a confirmed FLT3 ITD, TKD or ITD-F691L mutation documented within the past 90 days in absence of therapy or within the Screening period 28 days) prior to study drug administration on C1D1 if therapy has been given.
5. Patients must have previously been treated with Gilteritinib with failure to stop disease progression, or not met the criteria for treatment with Gilteritinib in the opinion of the Investigator, or chosen not to have treatment with Gilteritinib for social reasons.
6. Patients have a life expectancy of at least 3 months in the opinion of the Investigator.
7. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
8. Patient must meet the following criteria as indicated on the clinical laboratory tests:

   1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN)
   2. Serum total bilirubin ≤1.5 × ULN unless due to Gilbert's disease
   3. Estimated glomerular filtration (eGFR) rate of >50 mL/min as calculated by the Modification of Diet in Renal Disease equation.
9. Female patients:

   1. If of non-childbearing potential i.e., surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 6 weeks before the Screening visit or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone (FSH) level consistent with postmenopausal status, per local laboratory guidelines), or
   2. If of childbearing potential, must:

   i. Have a negative serum pregnancy test at the Screening visit and urine pregnancy test on admission to the clinic on Day-1.

   ii. Agree not to attempt to become pregnant or donate ova from signing the consent form until at least 45 days after the last dose of study drug.

   iii. Agree to use adequate contraception (defined as use of a condom by the male partner combined with use of a highly effective method of contraception from Screening until at least 45 days after the last dose of study drug, if not exclusively in a same-sex relationship or abstinent as a committed lifestyle).
10. Male patients and their female spouse/partners who are of childbearing potential must agree to use highly effective contraception consisting of 2 forms of birth control (at least 1of which must be a barrier method) starting at Screening and continue throughout the study period and for 45 days after the final study drug administration. Male patient must not donate sperm starting at Screening and throughout the study period and for 45 days after the final study drug administration.

Exclusion criteria

1. Diagnosis of isolated myeloid sarcoma (meaning, patients must have blood or marrow involvement with AML)
2. Acute promyelocytic leukemia (FAB M3)
3. Active central nervous system (CNS) involvement by AML
4. Clinical signs/symptoms of leukostasis requiring urgent therapy
5. Known active infection with Human Immunodeficiency Virus (HIV), hepatitis B or hepatitis C. Patients with a history of positive serology for hepatitis B or C require a negative Polymerase chain reaction (PCR) test for virus to go onto therapy
6. Disseminated intravascular coagulopathy with active, unmanageable bleeding or signs of thrombosis.
7. Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent; if the half-life of the agent is unknown, patients must wait 1 week prior to first dose of study treatment. An investigational agent is one for which there is no approved indication by the local regulatory authority.
8. Systemic antineoplastic therapy within 5 half-lives or radiation therapy within 1 week prior to starting protocol with the exception of hydroxyurea, which is allowed to control white blood cell counts.
9. Female patients who are pregnant or lactating
10. Patients with psychological, familial, social, or geographic factors, other significant medical condition, laboratory abnormality that otherwise preclude them from giving informed consent, following the protocol, potentially hamper compliance with study treatment and follow-up or would confound the interpretation of the results of the study.
11. Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction with evidence of residual abnormalities within 6 months prior to enrollment (Troponin (regular or high sensitivity) leak alone not included if no residual dysfunction), New York Heart Association (NYHA) Class III or IV heart failure, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Patients with medical comorbidities that will preclude safety evaluation of the combination should not be enrolled.
12. Infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control in the opinion of the Investigator. Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of DLTs | From baseline to the End of Treatment (EOT) (Max 24 cycles, 28 days each)
  To determine the maximum tolerated dose or biologically effective dose of ZE46-0134 in adults with FLT3 and spliceosome mutated relapsed and refractory AML.

SECONDARY OUTCOMES:
Incidence of AE/SAE | From baseline to the EOT (Max 24 cycles, 28 days each)
Incidence of clinically significant abnormal laboratory results | From baseline to the EOT (Max 24 cycles, 28 days each)
Incidence of abnormal clinically significant ECG results | From baseline to the EOT (Max 24 cycles, 28 days each)
Number of patients with AEs of Grade ≥ 3 | From baseline to the EOT (Max 24 cycles, 28 days each)
Number of treatment-related deaths | From baseline to the EOT (Max 24 cycles, 28 days each)
  Number of deaths, deemed related to the study drug by the Investigator
Plasma Cmax | PK samples will be collected throughout Cycles 1 and 2 (28 days each)
  ZE46-0134 peak plasma concentration
Plasma Css | PK samples will be collected throughout Cycles 1 and 2 (28 days each)
  ZE46-0134 steady state plasma concentration
Plasma Cmin | PK samples will be collected throughout Cycles 1 and 2 (28 days each)
  Minimum ZE46-0134 plasma concentration reached during a dosing interval
Plasma AUC | PK samples will be collected throughout Cycles 1 and 2 (28 days each)
  Area under the ZE46-0134 plasma concentration-time curve during a dosing interval
Number of patients attaining any type of Complete Remission (CR, CRh, CRi) by Cycle 6 | Up to 6 cycles (168 days total)
Number of patients attaining CR by Cycle 6 | Up to 6 cycles (168 days total)
Number of patients attaining response (CR, CRh, CRi, MLFS) by Cycle 6 | Up to 6 cycles (168 days total)

OTHER OUTCOMES:
Proportion of patients who became FLT3 ITD and TKD undetectable | During 6 Cycles of treatment (28 days each)
Number of patients with Genomic or proteomic abnormalities | From baseline to the EOT (Max 24 cycles, 28 days each)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Grove, Prof, Principal Investigator — Linear Clinical Research
Locations (23):
- United States (12):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - University of Kansas, Lawrence, Kansas
  - University of Maryland, College Park, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (3):
  - The Alfred Hospital, Melbourne, Victoria
  - Eastern Health - Box Hill Hospital, Melbourne, Victoria
  - Linear Clinical Research Ltd, Perth, Western Australia
- South Korea (4):
  - Gachon University Gil Medical Center, Incheon, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
- Taiwan (4):
  - Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taichung Veterans General Hospital, Xitun